CLINICAL TRIAL: NCT06611280
Title: Deuterium Metabolic Imaging in People with Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: DMI in MS
Record Dates: First submitted 2024-09-03; First posted 2024-09-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MS group: People with relapse remitting multiple sclerosis
  Interventions: Other: No Interventions
- HC group: Healthy control participant who are age- and sex-matched to the MS group
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No delivered intervention.

SUMMARY:
The goal of this case-control study is to investigate glucose brain metabolism in people with multiple sclerosis and age- and sex-matched healthy controls. The main questions it aims to answer are:

* How does brain glucose metabolism in people with multiple sclerosis compare to age- and sex-matched healthy controls?
* How is the brain glucose metabolism of people with multiple sclerosis associated with disease severity?

Participants will come in for testing lasting approximately three hours and undergo deuterium metabolic imaging, physical function test, cognitive function test, and answer survey.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years.
* Definite Relapsing remitting multiple sclerosis diagnosis according to the most recent diagnostic criteria

Exclusion Criteria:

* Contraindications for MRI:

Pacemaker, neurostimulator or cholera implant. Metal foreign bodies such as fragments and irremovable piercings. Unsafe medical implants (safety of heart valves, hips and the like must be confirmed).

Claustrophobia. Largest circumference including arms > 160 cm

* Pregnancy
* Competing neurological, psychiatric, or systemic diseases including diabetes (except prior TIA, unspecific brain MRI findings, hypertension, atherosclerosis and hyperlipidemia/cholesterolemia which are allowed).
* Participating in other clinical trials with investigational medical products or drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study seeks to include people with relapsing remitting multiple sclerosis that are otherwise healthy and age- and sex-matched healthy control participants.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
lactate to glx ratio | 2 hours from enrollment to end of assessment
  Brain deuterium metabolic imaging determined lactate to glx ratio

SECONDARY OUTCOMES:
Six-minute walk test | 3 hours from enrollment to end of assessment
  Measure of walking capacity as meters walking in six minutes
25 meter walk test | 3 hours from enrollment to end of assessment
  Maximal and usual walking speed over 25 feet including a 3 m measurement
Six-spot-step-test | 3 hours from enrollment to end of assessment
  Fastes time to kick six block away from six markings on the floor approximatly 1 meter from another in a zig-zag patteren.
Handgrip strength | 3 hours from enrollment to end of assessment
  Handgrip dynamometry
5-sit-to-stand | 3 hours from enrollment to end of assessment
  Time to perform five sit to stand.
Processing speed - Selective reminding test | 3 hours from enrollment to end of assessment
  Symbol digit modality test, number of symbols translated in 90 s
Memory function - Symbol digit modality test | 3 hours from enrollment to end of assessment
  Symbol digit modality test
  * Short term memory
  * consistence short term memory
  * long-term memory
Glukose level | 3 hours from enrollment to end of assessment
  From blood sample
Lactat level | 3 hours from enrollment to end of assessment
  From blood sample
Glucose uptake | 2 hours from enrollment to end of assessment
  Brain deuterium metabolic imaging demined glucose uptake measured by glucose to DHO + glucose ratio
glucose to glx ratio | 2 hours from enrollment to end of assessment
  Brain deuterium metabolic imaging demined glucose to glx ratio
Clinical information on multiple sclerosis - Disease modifying treatment | 7 days from enrollment to end of assessment
  Information on current disease modifying treatment are exacted from the hospital patient record
Clinical information on multiple sclerosis - Time since diagnosis | 7 days from enrollment to end of assessment
  Information on time since diagnosis are exacted from the hospital patient record
Modified Fatigue Impact Scale | 7 days from enrollment to end of assessment
  A 29-item questionnaire measuring the impact of multiple sclerosis on the patient. With a minimum score of 29 and a maximum of 116, a higher score indicates a worse outcome.
Clinical information on multiple sclerosis - Expanded disability status score | 7 days from enrollment to end of assessment
  Information on expanded disability status score is exacted from the hospital patient record. The expanded disability status score is a physician rating of disease severity from 0-10 with a higher score indicating higher disability.
Multiple Sclerosis Impact Scale | 7 days from enrollment to end of assessment
  A 21-item questionnaire measuring the impact of multiple sclerosis on the patient. With a minimum score of 0 and a maximum of 84, a higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to the European Unions General Data Protection Regulation.